CLINICAL TRIAL: NCT00403377
Title: Investigation of a Behavioral Substitute for Sunbathing
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CDR0000499830; R21CA109670 (NIH); UMASS-MCC-H-12102 (Other: University of Massachusetts Medical School); UMASS-MCC-H-11924 (Other: University of Massachusetts Medical School)
Record Dates: First submitted 2006-11-21; First posted 2006-11-23 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Melanoma (Skin); Skin Cancer
Keywords: melanoma; basal cell carcinoma of the skin; squamous cell carcinoma of the skin
MeSH Terms: conditions — Melanoma; Skin Neoplasms; Carcinoma, Basal Cell | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Phase II include two arms. In the intervention arm, photographs are taken of the participants and they then receive sunscreen lotion and sunless tanning lotion and instructions and benefits for using both. Participants also receive an educational pamphlet regarding skin cancer.
  Interventions: Behavioral: Intervention
- Control (No Intervention): Phase II include two arms. In the control arm, a souvenir photograph is taken of the participants and they then receive product samples that are irrelevant to skin cancer risk reduction (e.g., skin moisturizer, hair gel, chewing gum). Participants also receive educational materials at the completion of the study.

INTERVENTIONS:
Behavioral: Intervention — In the intervention arm, photographs are taken of the participants and they then receive sunscreen lotion and sunless tanning lotion and instructions and benefits for using both. Participants also receive an educational pamphlet regarding skin cancer.
  Arms: Intervention

SUMMARY:
RATIONALE: Understanding why sunbathers use or don't use sunless tanning products may help doctors plan effective ways to prevent skin cancer caused by sunbathing.

PURPOSE: This phase I/II trial is studying attitudes about the use of sunless tanning products and how well sunless tanning products work as a substitute for sunbathing in healthy participants.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine participants' attitudes regarding the benefits and barriers to using sunless tanning products after having sampled them. (Phase I)
* Determine participants' opinions, suggestions, and preferences regarding use of sunless tanning products. (Phase I)
* Determine the validity and reliability of the Sunless Tanning Attitudes Survey.
* Determine time spent sunbathing in random beach-goers. (Phase II)

Secondary

* Determine sunburn frequency in random beach-goers. (Phase II)
* Determine the use of a sunless tanner in these participants. (Phase II)
* Determine sun protection use in these participants. (Phase II)
* Determine perceptions of sun protection, susceptibility to photoaging, benefits of sunbathing, and severity of photoaging. (Phase II)

OUTLINE: This is an open-label phase I study followed by a pilot, randomized, controlled phase II study.

* Phase I (focus group): Participants complete the Sunless Tanning Attitudes (STA) survey, Sun Behavior (SB) survey, and the Decisional Balance for Sun Exposure and Sun Protection Questionnaire. Participants who have used a sunless tanner in the past also complete the Sunless Tanner Users (STU) survey. Participants receive sunless tanning lotion and instructions for its use. Participants are instructed to use the sunless tanner for 2 weeks (≥ 3 applications). Participants then complete the STA, SB, and STU surveys and participate in a focus group.
* Phase II:Participants are stratified by beach location and randomized to 1 of 2 intervention arms.

  * Arm I: Participants complete surveys as in phase I. Photographs are taken of the participants and they then receive sunscreen lotion and sunless tanning lotion and instructions and benefits for using both. Participants also receive an educational pamphlet regarding skin cancer.
  * Arm II: Participants complete surveys as in phase I. A souvenir photograph is taken of the participants and they then receive product samples that are irrelevant to skin cancer risk reduction (e.g., skin moisturizer, hair gel, chewing gum). Participants also receive educational materials at the completion of the study.

In both arms, participants complete surveys again at 2 and 12 months.

PROJECTED ACCRUAL: A total of 330 participants will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Self-described sun bather (phase I)

  * Intentional sun exposure lasting ≥ 1 hour to get a tan (outside or via tanning salon) at least twice a month during the months of June to August of the prior year
  * Intends to continue tanning during the coming summer months
* Random beach-goer (phase II)

PATIENT CHARACTERISTICS:

* Female
* Must speak English
* Must be able to read at the 6th grade level
* No prior sunless tanning products (phase I)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2006-04; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Phase 1 PO: Attitudes regarding the benefits and barriers to using sunless tanning products after having sampled them | Baseline and Focus Group
  The goal of the initial developmental phase of the present study is to determine the acceptability of sunless tanning as a substitute for sunbathing. Using focus groups comprised of sunbathers given the opportunity to sample sunless tanning products, we will identify perceived barriers and benefits of sunless tanning products, develop motivational messages encouraging the use of sunless tanning products, and preview intervention materials.
Phase II PO: Effectiveness of a beach-based pilot intervention (sun exposure at 2-, and 12- months follow-up) | Baseline, 2-, and 12-months
  The intervention will include sun damage imaging, sun safety and sunless tanning education/instruction, and the provision of samples of both sunscreen and sunless tanning products. Feasibility of the intervention, measures, and follow-up procedures will be assessed. The primary outcome for effectiveness will be sun exposure at 2-, and 12- months follow-up and a questionnaire only control group will be employed for comparison.

SECONDARY OUTCOMES:
Phase 1 SO: The second goal of the initial developmental phase will be to develop psychometrically sound measures of sunless tanner attitudes | Baseline and Focus Group
  To achieve this aim, psychometric analyses including inter-item analyses, autocorrelations, internal consistency, convergent and divergent validity will be conducted, and survey items will be added/revised (if necessary) based on content of focus group discussions.
Phase II SO: Sunburn frequency in random beach goers at 2 and 12 months | Baseline, 2-, and 12-months
  The intervention will include sun damage imaging, sun safety and sunless tanning education/instruction, and the provision of samples of both sunscreen and sunless tanning products. Feasibility of the intervention, measures, and follow-up procedures will be assessed. Secondary outcomes will include frequency of sunburns, use of sunless tanning products, sun protection behavior, and perceived benefits/barriers to sunbathing/sun protection.

CONTACTS AND LOCATIONS:
Overall Officials: Sherry L. Pagoto, PhD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

REFERENCES:
- [Result] Pagoto SL, Schneider KL, Oleski J, Bodenlos JS, Merriam P, Ma Y. Design and methods for a cluster randomized trial of the Sunless Study: a skin cancer prevention intervention promoting sunless tanning among beach visitors. BMC Public Health. 2009 Feb 5;9:50. doi: 10.1186/1471-2458-9-50. PMID 19196482
- [Derived] Pagoto SL, Schneider KL, Oleski J, Bodenlos JS, Ma Y. The sunless study: a beach randomized trial of a skin cancer prevention intervention promoting sunless tanning. Arch Dermatol. 2010 Sep;146(9):979-84. doi: 10.1001/archdermatol.2010.203. PMID 20855696